CLINICAL TRIAL: NCT04803851
Title: Anlotinib Plus Anti-PD-1 Antibody AK105 as Third or More-line Therapy for Advanced Pancreatic Cancer: a Prospective, Single-arm, Open-label, Pilot Study
Brief Title: Anlotinib Plus Anti-PD-1 Antibody AK105 for Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS2791
Record Dates: First submitted 2021-02-23; First posted 2021-03-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-02

CONDITIONS: Anlotinib; Anti-PD-1 Antibody; Advanced Pancreatic Cancer
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Anlotinib plus AK105
  Interventions: Drug: Anlotinib plus AK105

INTERVENTIONS:
Drug: Anlotinib plus AK105 — Anlotinib： a multi-kinase inhibitor AK105： an anti-PD-1 antibody

SUMMARY:
This study was designed to explore the clinical efficacy of Anlotinib combined with Anti-PD-1 antibody AK105 in the treatment of third- and above -line advanced pancreatic cancer patients, in order to find a better therapy strategy for pancreatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced or metastatic pancreatic cancer (PC),
* histologically or cytologically proven diagnosis of adenocarcinoma or adenosquamous carcinoma,
* failed to second-line chemotherapy for PC,
* 18-75 years of age,
* an Eastern Cooperative Oncology Group performance status score of 0 to 1,
* adequate organ functions

Exclusion Criteria:

* had received PD 1 /CTLA 4 antibody treatment
* had received anti-VEGFR inhibitors or antibodies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-06-29 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) based on RECIST v. 1 1 | 6 weeks
  Disease control rate (DCR) based on RECIST v. 1 1 by investigators

SECONDARY OUTCOMES:
Objective response rate (ORR) based on RECIST V. 1.1 | 6 weeks
  Objective response rate (ORR) based on RECIST V. 1.1 by investigators
Progression free survival (PFS) measured from the date of anlotinib plus AK105 initiation to the time of progression | 6 weeks
  Progression free survival (PFS) measured from the date of anlotinib plus AK105 initiation to the time of progression by investigators assessment
Overall survival (OS) measured from the date of anlotinib plus AK105 initiation to the time of death of any cause | 6 weeks
  Overall survival (OS) measured from the date of anlotinib plus AK105 initiation to the time of death of any cause by investigators assessment
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 weeks
  adverse events assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No